CLINICAL TRIAL: NCT04780490
Title: Comparison of the Effects of Perioperative Liberal and Restrictive Fluid Management on the Endothelial Glycocalyx Layer in Radical Cystectomy and Urinary Diversion
Brief Title: Comparison of Liberal and Restrictive Fluid Management on the Endothelial Glycocalyx in Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Associate Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018/374
Record Dates: First submitted 2020-02-06; First posted 2021-03-03 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Fluid Retention Tissue
Keywords: peroperative fluid management; restrictive fluid therapy; endothelial glycocalyx; Liberal fluid therapy
MeSH Terms: conditions — Edema

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- liberal fluid therapy (Active Comparator): Patients will be applied 2 mg midazolam for premedication. Before anesthesia induction, epidural catheter will be inserted to all patients and test dose will be made with 3 cc % 2 lidocaine (No medication from the epidural catheter will be administered during surgery).
  Standard anesthesia induction will be applied (fentanyl 2 mcg/kg; propofol 2 mg/kg; rocuronium 0.6 mg/kg ), and after intubation maintenance of anesthesia will be achieved with sevoflurane with a minimum alveolar concentration (MAC) of 0.8-1.
  Fluid resuscitation will be started with 10 ml / kg / hr Ringer's lactate solution.
  In patients with MAP <65 mmHg, 250 ml of Ringer's lactate solution will be given as a bolus.
  If the hypotension persists, the bolus 250 ml Ringer's lactate solution will be repeated up to 10 times.
  Interventions: Other: liberal fluid management
- restrictive fluid therapy (Active Comparator): Patients will be applied 2 mg midazolam for premedication. Before anesthesia induction, epidural catheter will be inserted to all patients and test dose will be made with 3 cc % 2 lidocaine ( No medication from the epidural catheter will be administered during surgery. ) Standard anesthesia induction will be applied ( fentanyl 2 mcg/kg; propofol 2 mg/kg; rocuronium 0.6 mg/kg ) and after intubation maintenance of anesthesia will be achieved with sevoflurane with a minimum alveolar concentration (MAC) of 0.8-1.
  Fluid resuscitation will be started with 2 ml / kg / hr Ringer's lactate solution and norepinephrine infusion at a dose of 2 mcg / kg / hr.
  In patients with MAP<65 mmHg, norepinephrine dose will be increased up to 8 mcg / kg / hr.
  If the hypotension persists although the norepinephrine dose is 8 mcg / kg / hr, 250 ml bolus Ringer's lactate solution will be given.
  Interventions: Other: restrictive fluid management

INTERVENTIONS:
Other: liberal fluid management — 10 ml/ kg/ hr Ringer's lactate solution
  Arms: liberal fluid therapy
Other: restrictive fluid management — 2 ml/ kg/ hr Ringer's lactate solution with 2 mcg / kg / hr norepinephrine infusion
  Arms: restrictive fluid therapy

SUMMARY:
The aim of this study is to compare the effect of the liberal and restrictive fluid treatments which are routinely performed in major urological surgeries in the perioperative period on ANP release and the endothelial glycocalyx layer.

In the study, the investigators aimed to compare changes in the glycocalyx structure by measuring the blood levels of ANP and heparan sulfate, hyaluronan and syndecan 1, which form the glycocalyx structure on the patients who received the liberal and restrictive fluid treatments during major urological surgeries.

DETAILED DESCRIPTION:
There is no strong evidence about the optimal fluid resuscitation for the patients undergoing major surgeries. Avoiding excess fluid resuscitation in the perioperative period is essential for reducing postoperative complications, morbidity and long-term mortality. In the perioperative period, ANP is released with increased wall stress in the cardiac atrium due to excess fluid loading. With the release of ANP, damage occurs in the glycocalyx layer, which is the structure primarily responsible for the permeability in the vascular endothelium.

Thus, the amount of ANP released from atrium and heparan sulfate, syndecan 1, hyaluronan in the glycocalyx layer structure increases in the blood.

The aim of this study is to compare changes in the glycocalyx structure by measuring the blood levels of ANP and heparan sulfate, hyaluronan and syndecan 1, which form the glycocalyx structure on the patients who received the liberal and restrictive fluid treatments during major urological surgeries. The blood samples will be taken at the beginning and at the end of the surgery.

The primary outcome of this study is the increase in ANP levels and heparan sulfate , hyaluronic acid, syndecan 1 levels which are the glycocalyx damage products in blood.

Secondary outcomes are intraoperative advanced hemodynamic cardiac measurement values, the amount of blood and blood products replaced to patients, duration of intensive care stay, duration of hospital stay, cardiac and respiratory complications, gastrointestinal complications, urinary complications, surgical complications such as anastomotic leaks, wound infection and fistula.

ELIGIBILITY:
Inclusion Criteria:

* ASA (The American Society of Anesthesiologists) status I-II-III patients
* Cases undergoing major urological surgery
* Cases for invasive artery monitoring and central venous catheterization
* Patients receiving general anesthesia
* Volunteering to participate in the study

Exclusion Criteria:

* Coagulopathy
* Patients with severe heart, kidney and liver dysfunction (EF <35% and / or GFR <30, Cre:> 2.5 and / or impaired liver function tests)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Atrial Natriuretic Peptide (ANP)( pg/mL) | The blood sample will be taken at beginning and end of the surgery
  Blood ANP concentration will be determined using an enzyme-linked immunosorbent assay kit
Heparan sulfate (ng/L) | The blood sample will be taken at beginning and end of the surgery
  Blood Heparan sulfate concentration will determine using an enzyme-linked immunosorbent assay kit
Syndecan 1 (pg/mL) | The blood sample will be taken at beginning and end of the surgery
  Blood Syndecan 1 concentration will be determined using an enzyme-linked immunosorbent
Hyaluronan (ng/L) | The blood sample will be taken at beginning and end of the surgery
  Blood Hyaluronan concentration will be determined using an enzyme-linked immunosorbent

SECONDARY OUTCOMES:
Amount of blood transfusion (unit) | From the beginning surgery to day 2 postoperatively
  Including red cell, fresh frozen plasma
Total intensive care unit (ICU) stay (Hour, day) | 30 days postoperative
  Including initial ICU admission and readmission times
Hospital stay (Hour, day) | 90 days postoperative
  From the beginning of surgery until actual hospital discharge
Gastrointestinal complications | 30 days postoperative
  Ileus, constipation, gastrointestinal bleeding, gastric ulcer, anastomotic intestinal leakage
Infectious complications | 30 days postoperative
  Urinary tract infection, pyelonephritis, urosepsis, pneumonia, wound infection
Surgical site complications | 30 days postoperative
  Wound dehiscence, evisceration
Genitourinary complications | 30 days postoperative
  Acute kidney injury, urethral anastamosis leak
Cardiac complications | 30 days postoperative
  Acute myocardial infarction, congestive heart failure, arrhythmia
Thromboembolic complications | 30 days postoperative
  pulmonary embolism
Stroke Volume Variation (SVV)(%) | From onset of the surgery up to end of the surgery, every 30 minutes
  SVV will be measured with Flo-Trac system (Edward Life Sciences). Normal range is about %10-15
Cardiac Index(CI )(l min-1 m-2), | From onset of the surgery up to end of the surgery, every 30 minutes
  CI will be measured with Flo-Trac system (Edward Life Sciences). Normal value is 2,6-4,2 l min-1 m-2
Systemic Vascular Resistance Index (SVRI )(dyn*s.cm-5 ) | From onset of the surgery up to end of the surgery, every 30 minutes
  SVRI will be measured with Flo-Trac system (Edward Life Sciences). Normal value is about 900-1300 dyn*s.cm-5

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Savran KARADENİZ, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

REFERENCES:
- See also: Restrictive deferred hydration combined with preemptive norepinephrine infusion during radical cystectomy reduces postoperative complications and hospitalization time: a randomized clinical trial. — https://www.ncbi.nlm.nih.gov/pubmed/23887199
- See also: Hypervolemia increases release of atrial natriuretic peptide and shedding of the endothelial glycocalyx. — https://www.ncbi.nlm.nih.gov/pubmed/25497357
- See also: Revised Starling equation and the glycocalyx model of transvascular ﬂuid exchange: an improved paradigm for prescribing intravenous ﬂuid therapy — https://www.ncbi.nlm.nih.gov/pubmed/22290457